CLINICAL TRIAL: NCT06212934
Title: "Chou's Tiaoshen" Acupoints for Short-term Insomnia: A Multicenter, Randomized, Controlled Clinical Study.
Brief Title: "Chou's Tiaoshen" Acupoints for Short-term Insomnia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li Huanqin, Chief physician, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYZD202203
Record Dates: First submitted 2023-12-22; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Short-term Insomnia
MeSH Terms: interventions — Acupuncture Therapy; Estazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Chou's Tiaoshen" acupoints group (Experimental): Acupuncturing"Chou's Tiaoshen" acupoints,"Chou's Tiaoshen" acupoints is derived from the experience of Zhou Dean, anational famous traditional Chinese medicine doctor in our department.
  Interventions: Other: Acupuncture
- Estazolam group (Active Comparator): Estazolam is a drug commonly used in the treatment of insomnia
  Interventions: Drug: Estazolam

INTERVENTIONS:
Other: Acupuncture — "Chou's Tiaoshen" acupoints includes Baihui (GV-20), Shenting (GV-24), and Sishencong (EX-HN1), Sanyinjiao (SP-6), Shenmen (HT-7) . Using stainless steel needles (0.32×40)mm, HuaTuo, China). Then some other points like, Danzhong(CV-17), Daling(PC-7), Taixi (KI-3), Qihai (CV-6), Taichong (LR3), and Qiuxu(GB-40) are chosen. Operation: Patients in supine position. Baihui (GV-20), Shenting (GV-24), and Sishencong (EX-HN1) are punctured at a depth of 20-25mm obliquely. Sanyinjiao (SP-6) and Shenmen (HT-7) are inserted 15mm perpendicularly. Until feeling tactile sensation then manually manipulated by rotation methods to produce a characteristic sensation known as "De Qi"; Technique: Mild reinforcing and attenuating, retaining the needle for 30minutes. The treatment will be givenonce a day and 5 times a week in weekdays, the course will last two weeks.
  Other Names: Dry needle
  Arms: "Chou's Tiaoshen" acupoints group
Drug: Estazolam — Participants will take estazolam 1mg 30min prior to bedtime everyday. The course of treatment is two weeks.
  Other Names: Estazolam pill
  Arms: Estazolam group

SUMMARY:
The goal of this clinical trial is to learn about the curative effect of "Chou's Tiaoshen" acupoints in short-term insomnia and the explore the possible mechanism of the action. The main questions it aims to answer are:

* Whether the curative effect of caupuncturing"Chou's Tiaoshen" acupoints in the treatment of short-term insomnia is not inferior to that of Esazolam.
* What is the possible mechanism of acupuncture "Chou's Tiaoshen"acupoints for short-term insomnia.

Participants with short-term insomnia who met the criteria will be randomly assigned to "Chou's Tiaoshen"acupoints group and Esazolam group. Polysomnography, heart rate variability, cortisol and related scales will be measured before and after treatment to detect the changes in symptoms and signs before and after treatment.

DETAILED DESCRIPTION:
The incidence of short-term insomnia is high. In clinical practice, due to patients insufficient understanding of the severity of short-term insomnia and the side effects of drug treatment, the treatment of short-term insomnia has not made breakthrough progress, and some patients may turn into chronic insomnia, which is more harmful. There is a growing consensus that short-term insomnia is a hyperarousal disorder associated with high sleep reactivity. "Chou's Tiaoshen" acupoints is derived from the experience of Zhou Dean, a national famous traditional Chinese medicine doctor in our department, and the main points are selected: Baihui (DU20), Shenting (DU24), Sishencong (EX-HN1), Shenmen (HT7), Neiguan (PC6), and Sanyinjiao (SP6), the acupuncture method has achieved good clinical efficacy in the early insomnia research, which can improve the waking state of insomnia patients during the day and improve the sleep quality at night. In order to further verify the efficacy of "Chou's Tiaoshen" acupoints in the treatment of short-term insomnia, explore the possible mechanism of action, discover the physical characteristics of patients with short-term insomnia, and explain the connotation of "Chou's Tiaoshen" acupoints, this clinical study is conducted. 96 patients with short-term insomnia who meet the inclusion criteria will be selected and divided into the "Chou's Tiaoshen" acupoints group and the oral esazolam group according to the principle of random allocation. The study will be conducted in the acupuncture and moxibustion Department of Beijing Hospital of Traditional Chinese Medicine and Shunyi Hospital of Beijing Hospital of Traditional Chinese Medicine. Pittsburgh Sleep Scale (PSQI) assessment, polysomnography (PSG, some subjects), heart rate variability (HRV) monitoring, serum cortisol measurement will be performed before and after treatment. Ford Insomnia Stress Response Test (FIRST) scale, Daytime function Scale and Chinese Medicine Symptom Score Scale will be evaluated to evaluate the efficacy and explore the mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Meet diagnostic criteria for short-term insomnia according to the Diagnostic and Statistical Manual of Mental Disorders Text Revision, 5th ed (DSM-V) and Chinese Adult Insomnia Diagnosis and Treatment Guide 2017，a predominant complaint of dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms: 1)Difficulty initiating sleep. 2). Difficulty maintaining sleep, characterized by frequent awakenings or problems returning to sleep after awakenings. 3)Early-morning awakening with inability to return to sleep. 4)The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning. The sleep difficulty occurs at least 3 nights per week. The duration of the sleep difficulty is 1 week to 3 months.
2. Experienced insomnia between 1 weeks and 3 months before the start of project.
3. Age: patients between 18 and 70 years old.
4. Patients who agreed to participant in this trial and assigned the informed consent.

Exclusion Criteria:

1. People with other DSM-IV Axis I, Axis II mental disorders or substance abuse/dependence;
2. Patients with serious primary diseases such as cardiovascular and cerebrovascular diseases, hypertension, digestive system, hematopoietic system, liver, kidney, or severe anxiety and depression;
3. Caused by alcohol or drugs;
4. Pregnant or lactating women;
5. Easy to combine infection and bleeding; 6.1 Patients who have used psychotropic drugs, such as antidepressants, mania drugs or other drugs used to treat psychosis, in the last month, and patients who have taken sleeping pills in the last 1 month;

7. Those who cannot cooperate with treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | PSQI will be recorded 3 times, before treatment, and at the 14th day , 28th day after treatment.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. Eighteen individual items generate seven "component" scores: subjective sleep quality (SQ), sleep-onset latency (SOL), total sleep time (TST), habitual sleep efficiency (SE), sleep disturbances ( Dyssomnia), use of sleeping medication, and daytime dysfunction (DD).The cumulative component score is the PSQI total score ranging from 0 to 21, higher scores indicates worse sleep quality.

SECONDARY OUTCOMES:
Polysomnography | PSG will be recorded in 10 randomly selected patients in each group before treatment and 14 days after treatment.
  Polysomnography (PSG) is a classic instrument for detecting sleep conditions.The following data can be obtained by PSG monitoring: total sleep time, sleep latency, The percentage of time spent in each sleep stage. PSG is of great value for the degree and differential diagnosis of insomnia.
Heart Rate Variability (HRV) | HRV will be recorded 3 times, before treatment, at the 14th day and 28th day after treatment.
  The degree and regularity of heart rate changes can be reflected by measuring the variability of continuous normal R-R interphase changes by dynamic elctrocardiogram, so as to judge its impact on cardiovascular activities, which can reflect the activity of autonomic nervous system and quantitatively evaluate the balance of sympathetic and vagal nerve tension.
Concentration of serum cortisol | Serum cortisol will be recorded 2 times, before treatment, and at the 14th day , 28th day after treatment, and the measurement time was fixed at 8 am each time.
  Serum cortisol is elevated during stress, which can reflect excessive arousal, and if the brain is constantly under high stress, may lead to long-term elevated cortisol levels.
Fatigue Scale | FS will be recorded 3 times, before treatment, and at the 14th day , 28th day after treatment.
  The fatigue scale(FS) consists of 14 items, each of which is a fatigue-related question, reflecting both physical fatigue and mental fatigue. The highest total score is 14 points, the lowest is 0 points, and the higher the score is, the more serious the fatigue is.
Ford Insomnia Response to Stress Test Chinese version，FIRST | FIRST will be recorded 3 times, before treatment, and at the 14th day , 28th day after treatment.
  FIRST is a self-reporting tool including nine items designed to assess sleep response, The minimum total score is 9 and the maximum is 36. Higher scores on the FIRST indicate a more highly reactive sleep system.
Traditional Chinese medicine symptom scoring Scale | TCM symptom score will be recorded 3 times, before treatment, and at the 14th day , 28th day after treatment.
  The TCM symptom scoring scale consists of five items with a minimum score of 0 and a maximum score of 30, reflecting the five core symptoms of insomnia, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Huanqin Li, Doctor, Study Chair — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish a protocol of this trial in about 6-8 months after the registration, and one paper of the trial including results in a high-impact peer reviewed journal in one year after the trial. About two years after the end of this trial and our open publication of the result, the primary data and type of analysis will be available for 5-10 years until data updated by a more specific study with larger number of participants. Anyone who are interested in the trial can ask us to share the primary data by send a requirement through email. We provide the collected primary data without no real information of participants, all the data sequence will be numbered instead of real names.
Supporting Information: Study Protocol, CSR
Time Frame: About two years after the end of this trial and our open publication of the result, the primary data and type of analysis will be available for 5-10 years until data updated by a more specific study with larger number of participants.
Access Criteria: Anyone who are interested in the trial can ask us to share the primary data by send a requirement through email.
URL: https://trialsjournal.biomedcentral.com/